CLINICAL TRIAL: NCT03858478
Title: Initiation of First-line Antiretroviral Treatment With TENOFOVIR ALAFENAMIDE - EMTRICITABINE - BICTEGRAVIR at the First Clinical Contact in France
Brief Title: Initiation of First-line Antiretroviral Treatment With TENOFOVIR ALAFENAMIDE - EMTRICITABINE - BICTEGRAVIR at the First Clinical Contact in France: Trial IMEA 055 - FAST
Acronym: FAST
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMEA 055- FAST
Record Dates: First submitted 2019-02-25; First posted 2019-02-28 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-11

CONDITIONS: HIV Seropositivity
Keywords: HIV, new diagnosis, Biktarvy
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Intervention Model Description: Pilot study, single arm, multicentric, national
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biktarvy arm (Experimental): one tablet of BIKTARVY including [TAF (25mg) / FTC (200mg) / BICTEGRAVIR (50mg) ] one tablet once a day for 48 weeks
  Interventions: Drug: Biktarvy arm

INTERVENTIONS:
Drug: Biktarvy arm — BIKTARVY : one tablet QD, every day between D0 and M12 includind - TAF (25mg) / FTC (200mg) / BICTEGRAVIR (50mg)

SUMMARY:
Evaluation of antiretroviral treatment adherence using determination of Bictegravir, Emtricitabine and Tenofovir with new HIV patients in France

DETAILED DESCRIPTION:
* Patient treated at the first clinical contact
* 18 sites (hospitals) in France
* Treatment during 48 weeks with principal objective at W24 (plasma HIV-RNA < 50 copies/ml)
* Evaluation of antiretroviral treatment adherence using determination of Bictegravir, Emtricitabine and Tenofovir in hair sample

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* newly diagnosed HIV-infected individual evidenced by any of the following tests: (i) positive self-test, (ii) positive HIV Rapid antibody test, (iii) positive HIV immunoassay (ELISA 4th generation) test
* antiretroviral-treatment naive
* negative urine pregnancy test for women of childbearing potential and willing to use effective contraception (mechanical or medicamental)
* willing to sign an informed written consent-
* regular health insurance
* willing to provide two distinct contact information (telephone number and/or email) in order to be easily reached if needed between Day 0 and Day 7

Exclusion Criteria:

* clinical symptoms suggestive of opportunistic infections
* participant not willing to provide two distinct contact information
* a woman who is pregnant or breast-feeding or planning to become pregnant during the expected study period.
* Co-medication with deleterious interaction with study treatment (eg enzyme inducer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
To achieve virological suppression (plasma HIV-RNA < 50 copies/ml) at Month 6 (M6)on study treatment with a first-line treatment with TAF / FTC/ BIC initiated at the first clinical contact (Snapshot method) | virological suppression at Month 6 (M6)

SECONDARY OUTCOMES:
proportion of participants with a false positive HIV screening test (i.e. a first positive test that has not been confirmed) | DAY 0 (D0)
proportion of participants with plasma HIV-RNA < 50 copies/ml | Month 1 (M1), Month 3 (M3), Month 6 (M6), Month 9 (M9), Month 12 (M12)
change in CD4 T cell count | between DAY 0 (D0) and Month 3 (M3), Month 6 (M6) and Month 12 (M12)
change in CD4/CD8 ratio | between DAY 0 (D0) and Month 6 (M6) and Month 12 (M12)
proportion of participants requiring discontinuation/modification of TAF/FTC/Bictegravir due to (i) Baseline resistance to one of the study drugs, (ii) adverse events leading to study treatment discontinuation/Modification | Between DAY 0 (D0) and Month 12 (M12)
proportion of participants experiencing a grade 3-4 adverse event (related or not related to study treatment) | Between DAY 0 (D0) and Month 12 (M12)
proportion of participants with protocol defined virological failure (plasma HIV-RNA > 400 copies/ml at Week 12 confirmed on a second sample drawn 15-21 days later, or two consecutive plasma HIV-RNA > 50 copies/ml within 15-21 days as of Week 24) | Between Month 6 (M6) and Month 12 (M12)
proportion of participants harboring a virus developing resistance-associated mutations at the time of protocol-defined virological failure | Between Month 6 (M6) and Month 12 (M12)
number of comedications used during the 12-months study period | Between DAY 0 (D0) and Month 12 (M12)
adherence to study treatment evaluated by drug concentrations measurement in hair | Month 1 (M1), Month 3 (M3), Month 6 (M6) and Month 12 (M12)
proportion of participants lost to follow-up throughout the 12-months study period (LFU = having missed more than two consecutive visits except for W24 and W48 visit) | Between DAY 0 (D0) and Month 12 (M12)
participants' acceptability of immediate antiretroviral initiation treatment (self-assessed auto-questionnaires | At Day 0 (D0), Month 3 (M3), Month 6 (M6) and Month 12 (M12)
adherence to study treatment evaluated by (i) self-assessed auto-questionnaires (4-day recall), | Month 1 (M1), Month 3 (M3), Month 6 (M6) and Month 12 (M12)
adherence to study treatment evaluated by drug concentrations measurement in plasma | Month 1 (M1), Month 3 (M3), Month 6 (M6) and Month 12 (M12)
type of comedications used during the 12-months study period | Between DAY 0 (D0) and Month 12 (M12)

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Hopital Zobda Quitman, Fort-de-france, Martinique
  - Hôpital Pellegrin - Service de Médecine Interne et Maladies Infectieuses, Bordeaux
  - Hôpital Côte de Nacre - Service des Maladies Infectieuses, Caen
  - Centre hospitalier Sud Francilien, Corbeil-Essonnes
  - Hôpital Henri Mondor - Service d'Immunologie Clinique, Créteil
  - Hopital Francois Mitterrand, Dijon
  - Hopital Raymond Poincare, Garches
  - Hopital Sainte-Marguerite, Marseille
  - Hôpital Gui de Chauliac - Service de Maladies Infectieuses et Tropicales, Montpellier
  - L'ARCHET, Nice
  - Hopital Saint Antoine, Paris
  - Hopital Necker, Paris
  - Hopital Bichat, Paris
  - Hopital Tenon, Paris
  - Hopital Foch, Suresnes
  - Hopital Gustave Dron, Tourcoing
  - Hopital Bretonneau, Tours